CLINICAL TRIAL: NCT04246021
Title: The Use of Intravenous Ferric Carboxymaltose (FCM) Without Erythropoiesis-stimulating Agents (ESA) in the Treatment of Anemia in Cancer Patients Undergoing Chemotherapy With or Without Radiotherapy
Brief Title: Use of Intravenous Ferric Carboxymaltose in Treatment of Anemia in Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Hussein Cancer Center (Other)
Collaborators: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Principal Investigator, Hikmat Abdel-Razeq, Chief Medical Officer and Deputy Director General King Hussein Cancer Center, King Hussein Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRT-INM-0615/09
Record Dates: First submitted 2020-01-26; First posted 2020-01-29 (Actual); Results first posted 2021-12-08 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Anemia; Cancer
MeSH Terms: conditions — Anemia; Neoplasms | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: This study is a nonrandomized, single arm, open-label study stratified by iron-deficiency status.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferric carboxymaltose (ferrinject) (Experimental): Patients will receive one or two doses of Ferric carboxymaltose (ferrinject), based on the body weight and Hb level.
  * Ferric carboxymaltose will be administered as a single infusion if the needed dose is 1000 mg as a short IV infusion
  * If the needed Ferric carboxymaltose dose is > 1000 mg, an initial dose of 1000 mg will be given as a short IV infusion and the remaining dose will be given the week after in a similar fashion
  Interventions: Drug: Ferric carboxymaltose (FCM)

INTERVENTIONS:
Drug: Ferric carboxymaltose (FCM) — intravenous iron formulation
  Other Names: Ferinject

SUMMARY:
This study is a nonrandomized, single arm, open-label study stratified by iron-deficiency status.

DETAILED DESCRIPTION:
The study aims to investigate the effect of FCM (without ESAs) on anemic cancer patients undergoing chemotherapy (with or without radiotherapy); stratified by status of iron deficiency (i.e. non-iron deficient vs. iron deficient patients ). The study will also try to find out whether serum level of Hepcidin and C reactive protein can correlate with response

Patients will receive one or two doses of FCM, based on the body weight and Hb level. Patients will be followed-up for a total of twelve weeks. The study is divided into a screening, treatment and follow-up phases and is expected to be completed in 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult more than or equal 18 years old at the time of informed consent.
* Patient has pathologic diagnosis of solid tumor (breast cancer, colorectal, lung, sarcoma, head and neck, sarcoma, genitourinary or gynecological cancer).
* Patients who started chemotherapy (with or without radiotherapy) or planned to receive chemotherapy for at least 12 weeks.
* Patient has an Eastern Cooperative Oncology Group performance status between 0 and 2.
* Patient with Hb ≤11 g/dL.
* Patient has a Life expectancy at least 6 months.
* Adequate hepatic and renal function defined as a serum aspartate aminotransferase or alanine aminotransferase level that are no more than 3 times the upper limit of the normal range, a serum bilirubin level that is no more than 2 times the upper limit of the normal range and a serum Creatinine level of less than 2 mg per deciliter.
* Patient is able to understand and provide informed consent to participate in the study.

Exclusion Criteria:

* Patient has Hb < 8.0 g/dL
* Patient presenting with hematologic malignancy including
* Prior gastric surgery.
* Patients on definitive radiotherapy alone.
* Patients with relevant history (within six weeks) or clinical evidence of hemolysis or active bleeding that could, in the investigator's judgment, be a potential cause for the anemia (no gross hematuria, hemoptysis, hematochezia or melena and negative stool for hemoccult)
* Presence of other nutritional anemia; deficiency of vitamin B12 less than 187 pg/ml and deficiency of Folate less than 3.1 ng/ml according to the local laboratory normal ranges
* Patient has Iron overload (Serum Ferritin more than 800 ng/ml or Transferrin saturation (TSAT) more than 40%)
* Patient is pregnant or lactating.
* Patient has a personal or family history of hemochromatosis.
* Patient has hypersensitivity to any form of IV iron.
* Patient has received red blood cells transfusion or used erythropoietin within 2 weeks of enrollment into the study.
* Patient has received any form of intravenous iron within the last 12 weeks
* Patient has received oral iron supplements within 1 month of enrollment to the study, except for multivitamin supplements containing less than 30 mg iron.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Razeq H, Saadeh SS, Malhis R, Yasser S, Abdulelah H, Eljaber R, Kleib A, Ismael R. Treatment of anemia in cancer patients undergoing chemotherapy with intravenous ferric carboxymaltose without erythropoiesis-stimulating agents. Ther Adv Med Oncol. 2020 Sep 9;12:1758835920953292. doi: 10.1177/1758835920953292. eCollection 2020. PMID 32952616

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferric Carboxymaltose (Ferrinject): Patients will receive one or two doses of Ferric carboxymaltose (ferrinject), based on the body weight and Hb level.
  * Ferric carboxymaltose will be administered as a single infusion if the needed dose is 1000 mg as a short IV infusion
  * If the needed Ferric carboxymaltose dose is > 1000 mg, an initial dose of 1000 mg will be given as a short IV infusion and the remaining dose will be given the week after in a similar fashion
  Ferric carboxymaltose (FCM): intravenous iron formulation
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (Ferrinject)
Started | 84
Completed | 84
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 84 adult cancer patients on active chemotherapy with hemoglobin (Hb) level ⩽11.0 g/dL were recruited.
  Based on serum ferritin (sFr) and transferrin saturation(TSAT), patients were divided into 3 groups: group I (absolute iron deficiency, n = 26) with sFr < 30 ng/mL and TSAT < 20%; group II (functional iron deficiency, n = 24) with sFr 30-800 ng/mL and TSAT < 20%; and patients with TSAT ⩾ 20% were placed in group III as "others" (n = 34).
Arm/Group | Ferric Carboxymaltose (Ferrinject)
Number analyzed (Participants) | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Jordan | 84

OUTCOME MEASURES:

1. Primary Outcome: The Median Hb Change From Baseline to Week 12
Description: The median Hb change from baseline to week 12 per patient in the three groups, Based on serum ferritin (sFr) and transferrin saturation(TSAT), patients were divided into the 3 groups: group I (absolute iron deficiency, n = 26) with sFr < 30 ng/mL and TSAT < 20%; group II (functional iron deficiency, n = 24) with sFr 30-800 ng/mL and TSAT < 20%; and patients with TSAT ⩾ 20% were placed in group III as "others" (n = 34).
Time Frame: up to 12 weeks
Population: median Hb change from baseline to week 12
Measure: Median (Full Range); unit: gm/dl
Groups:
- Ferric Carboxymaltose (Ferinject) in Patients With Absolute Iron Deficiency Anemia; Ferric Carboxymaltose (Ferinject) in Patients With Functional Iron Deficiency; Others-Ferric Carboxymaltose(Ferinject) in Patients With Anemia: A total of 84 adult cancer patients on active chemotherapy with hemoglobin (Hb) level ⩽11.0 g/dL were recruited.
  Based on serum ferritin (sFr) and transferrin saturation(TSAT), patients were divided into 3 groups: group I (absolute iron deficiency, n = 26) with sFr < 30 ng/mL and TSAT < 20%; group II (functional iron deficiency, n = 24) with sFr 30-800 ng/mL and TSAT < 20%; and patients with TSAT ⩾ 20% were placed in group III as "others" (n = 34).
Arm/Group | Ferric Carboxymaltose (Ferinject) in Patients With Absolute Iron Deficiency Anemia | Ferric Carboxymaltose (Ferinject) in Patients With Functional Iron Deficiency | Others-Ferric Carboxymaltose(Ferinject) in Patients With Anemia
Number analyzed (Participants) | 26 | 24 | 34
gm/dl | 2.35 [-1 to 4.6] | 1.5 [-1 to 3.7] | 0.5 [-1.6 to 3.3]

2. Primary Outcome: Percentage of Patients With Hb Increment of at Least 1.0 gm/dL.
Description: Percentage of patients with Hb increment of at least 1.0 gm/dL during their participation (from baseline to week 12 per patient) in the three groups,
  Based on serum ferritin (sFr) and transferrin saturation(TSAT), patients were divided into the 3 groups: group I (absolute iron deficiency, n = 26) with sFr < 30 ng/mL and TSAT < 20%; group II (functional iron deficiency, n = 24) with sFr 30-800 ng/mL and TSAT < 20%; and patients with TSAT ⩾ 20% were placed in group III as "others" (n = 34).
Time Frame: up to 12 weeks
Population: Response defined as a Hb increment ⩾1.0gm/dL
Measure: Count of Participants; unit: Participants
Groups:
- Ferric Carboxymaltose (Ferinject) in Patients With Absolute Iron Deficiency Anemia; Ferric Carboxymaltose (Ferinject) in Patients With Functional Iron Deficiency; Others-Ferric Carboxymaltose(Ferinject) in Patients With Anemia: Based on serum ferritin (sFr) and transferrin saturation(TSAT), patients were divided into 3 groups: group I (absolute iron deficiency, n = 26) with sFr < 30 ng/mL and TSAT < 20%; group II (functional iron deficiency, n = 24) with sFr 30-800 ng/mL and TSAT < 20%; and patients with TSAT ⩾ 20% were placed in group III as "others" (n = 34).
Arm/Group | Ferric Carboxymaltose (Ferinject) in Patients With Absolute Iron Deficiency Anemia | Ferric Carboxymaltose (Ferinject) in Patients With Functional Iron Deficiency | Others-Ferric Carboxymaltose(Ferinject) in Patients With Anemia
Number analyzed (Participants) | 26 | 24 | 34
Participants | 21 | 17 | 12

3. Primary Outcome: Percentage of Patients Achieving Correction of Anemia (Hb >11.0 gm/dL)
Description: Percentage of patients achieving correction of anemia (Hb >11.0 gm/dL) during their participation (from baseline to week 12 per patient) in the three groups.
  A total of 84 adult cancer patients on active chemotherapy with hemoglobin (Hb) level ⩽11.0 g/dL were recruited.
  Based on serum ferritin (sFr) and transferrin saturation(TSAT), patients were divided into 3 groups: group I (absolute iron deficiency, n = 26) with sFr < 30 ng/mL and TSAT < 20%; group II (functional iron deficiency, n = 24) with sFr 30-800 ng/mL and TSAT < 20%; and patients with TSAT ⩾ 20% were placed in group III as "others" (n = 34).
Time Frame: up to 12 weeks
Population: count of patients achieving correction of anemia
Measure: Count of Participants; unit: Participants
Groups:
- Others, Ferric Carboxymaltose(Ferinject) in Patients With Anemia: A total of 84 adult cancer patients on active chemotherapy with hemoglobin (Hb) level ⩽11.0 g/dL were recruited.
  Based on serum ferritin (sFr) and transferrin saturation(TSAT), patients were divided into 3 groups: group I (absolute iron deficiency, n = 26) with sFr < 30 ng/mL and TSAT < 20%; group II (functional iron deficiency, n = 24) with sFr 30-800 ng/mL and TSAT < 20%; and patients with TSAT ⩾ 20% were placed in group III as "others" (n = 34).
Arm/Group | Ferric Carboxymaltose (Ferinject) in Patients With Absolute Iron Deficiency Anemia | Ferric Carboxymaltose (Ferinject) in Patients With Functional Iron Deficiency | Others, Ferric Carboxymaltose(Ferinject) in Patients With Anemia
Number analyzed (Participants) | 26 | 24 | 34
Participants | 20 | 17 | 18

4. Secondary Outcome: Response Rate in Relation to Baseline Iron Deficiency Status
Description: Response rate in relation to baseline iron deficiency status; Patients were considered responders if they showed a minimum of 1.0 gm/dL increment in Hb level during their participation (from baseline to week 12 per patient)
  Based on serum ferritin (sFr) and transferrin saturation(TSAT), patients were divided into 3 groups: group I (absolute iron deficiency, n = 26) with sFr < 30 ng/mL and TSAT < 20%; group II (functional iron deficiency, n = 24) with sFr 30-800 ng/mL and TSAT < 20%; and patients with TSAT ⩾ 20% were placed in group III as "others" (n = 34).
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Others, Ferric Carboxymaltose(Ferinject) in Patients With Anemia: Based on serum ferritin (sFr) and transferrin saturation(TSAT), patients were divided into 3 groups: group I (absolute iron deficiency, n = 26) with sFr < 30 ng/mL and TSAT < 20%; group II (functional iron deficiency, n = 24) with sFr 30-800 ng/mL and TSAT < 20%; and patients with TSAT ⩾ 20% were placed in group III as "others" (n = 34).
Arm/Group | Ferric Carboxymaltose (Ferinject) in Patients With Absolute Iron Deficiency Anemia | Ferric Carboxymaltose (Ferinject) in Patients With Functional Iron Deficiency | Others, Ferric Carboxymaltose(Ferinject) in Patients With Anemia
Number analyzed (Participants) | 26 | 24 | 34
Participants | 21 | 17 | 12

5. Secondary Outcome: Percentage of Patients Who Will Require Blood Transfusion or ESA Treatment
Description: Percentage of patients who received red blood cells (RBCs) transfusion or used erythropoietin during their participation (from baseline to week 12 per patient) among the 84 recruited adult cancer patients on active chemotherapy with hemoglobin (Hb) level ⩽11.0 g/dL
Time Frame: up to 12 weeks
Population: Percentage of patients who will require blood transfusion or ESA treatment
Measure: Count of Participants; unit: Participants
Groups:
- Ferric Carboxymaltose (Ferrinject): Percentage of patients who received red blood cells (RBCs) transfusion or used erythropoietin during their participation (from baseline to week 12 per patient) among the 84 recruited adult cancer patients on active chemotherapy with hemoglobin (Hb) level ⩽11.0 g/dL
Arm/Group | Ferric Carboxymaltose (Ferrinject)
Number analyzed (Participants) | 84
Participants | 6

ADVERSE EVENTS:
Time Frame: up to 12 weeks from drug administration
Arm/Group | Ferric Carboxymaltose (Ferinject) in Patients With Absolute Iron Deficiency Anemia | Ferric Carboxymaltose (Ferinject) in Patients With Functional Iron Deficiency | Others-Ferric Carboxymaltose(Ferinject) in Patients With Anemia
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/34
Other Adverse Events (participants affected / at risk) | 17/26 | 6/24 | 16/34
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (Ferinject) in Patients With Absolute Iron Deficiency Anemia (N=26) | Ferric Carboxymaltose (Ferinject) in Patients With Functional Iron Deficiency (N=24) | Others-Ferric Carboxymaltose(Ferinject) in Patients With Anemia (N=34)
hypophosphatemia (Investigations) | 17 | 6 | 16 — hypophosphatemia

LIMITATIONS AND CAVEATS:
study population is small, and some caution is required before generalizing study results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT04246021/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT04246021/SAP_001.pdf